CLINICAL TRIAL: NCT04389385
Title: Aerosol Inhalation of the Exosomes Derived From Allogenic COVID-19 T Cell in the Treatment of Early Stage Novel Coronavirus Pneumonia
Brief Title: COVID-19 Specific T Cell Derived Exosomes (CSTC-Exo)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Mustafa Cetin, Professor, TC Erciyes University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: EruCovid2020
Record Dates: First submitted 2020-05-12; First posted 2020-05-15 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Corona Virus Infection; Pneumonia
Keywords: Corona virus; COVID-19; Pnemonia; Cell therapy; Virus specific T cell; Exosome
MeSH Terms: conditions — Coronavirus Infections; Pneumonia; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- COVID-19 STCs -Exo therapy (Experimental): In addition to the best available treatment, participants will receive inhaler COVID-19 STCs -Exo therapy *.
  Biological: Inhaler CSTH-Exo treatment will be applied daily x 5 times (2.0 x 108 nano vesicle / 3 ml; on day 1 to day 5).
  * If the improvement contribution is observed in the parameters, this application period could be extended
  Interventions: Biological: COVID-19 Specific T Cell derived exosomes (CSTC-Exo)

INTERVENTIONS:
Biological: COVID-19 Specific T Cell derived exosomes (CSTC-Exo) — The virus-specific T-cells (VSTs) are body's natural immune defense against various disease-causing viruses. Donor originated COVID-19 specific T-cells (CSTC) are in vitro activated and expanded by exposing to viral peptide fragments in the presence of natural immune stimulant proteins called cytokines. These Covid-19 specific fragment peptides activate specific T-cells and stimulate the secretion of potent mediators including IFN gamma in forms of exosomes. We propose treatment of Covid-19 patients -who are at early stages of pulmonary disease- with CSTC-exomes to control disease progression.

SUMMARY:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) pandemic has caused mass mortality in the last 3 months that necessitates urgent development of new therapeutical agents. So far there is no effective anti-viral drug to reduce viral load that has critical importance to prevent progress into severe viral pneumonia and systemic hyper inflammation state. This project is to offer a biologic agent based on T cell derived exosomes. This is a novel approach using our proprietary protocols for drug development. This clinical trial is to test the safety and efficacy of this new agent following targeted delivery by metered dose inhaler. The project have received proper approvals from the Turkish Ministry of Health and Erciyes University, Kayseri Turkey. Turk-Patent Application Number: PCT/TR2020/050302

DETAILED DESCRIPTION:
The Covid-19 disease due to infection with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) has affected millions people and caused thousands of mortality in the world over the last 3 months. Clinically, COVID-19 presents with a wide range of disease severity ranging from asymptomatic or very mild flu-like symptoms to very severe acute respiratory syndrome and multi-organ failure. The severity of COVID-19 correlates with escalating levels of systemic inflammation that eventually leads to hyperinflammatory stage resembling macrophage activation syndrome and death. Therefore, early intervention is essential to prevent progress into respiratory failure that requires reduction of viral load.

The virus-specific T-cells (VSTs) are body's natural immune defense against various disease-causing viruses. Donor originated COVID-19 specific T-cells (CSTC) are in vitro activated and expanded by exposing to viral peptide fragments in the presence of natural immune stimulant proteins called cytokines. These COVID-19 specific fragment peptides activate specific T-cells and stimulate the secretion of potent mediators including IFN gamma in forms of exosomes. We propose treatment of COVID-19 patients -who are at early stages of pulmonary disease- with CSTC-exomes to control disease progression. This biological agent offers universal application without a need for HLA match. Furthermore, exosomes are suitable as "off the shelf product" that allows dose titration for personalized treatment.

The purpose of this single arm open labeled, combined interventional (phase I/II trials) clinical trial is to explore the safety and efficiency of inhaled CSTC-exomes in the treatment of early stage novel coronavirus (NCV) pneumonia.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness of study participant to accept this treatment arm, and signed informed consent;
2. Male or female, aged at 18 years (including) to 75 years old;
3. Confirmation of SARS-CoV-2 infection by reverse-transcription polymerase chain reaction (RT-PCR) from respiratory tract or blood specimens;
4. Patients with confirmed novel coronavirus pneumonia per imaging and clinical findings;
5. Diagnostic criteria of "Early Stage NCV Pneumonia " includes:

   1. Respiratory rate (RR) ≥ 30 times/min
   2. Pulse oxygen saturation (SpO2) at rest ≤ 93%
   3. Oxygenation Index: (PaO2/FiO2: ≥ 100mmHg and ≤ 300mmHg)

Exclusion Criteria:

1. The patients showing finding of late severe pneumonia (PaO2/FiO2: < 100mmHg) with systemic hyperinflammation, shock, and multi organ involvement
2. Allergic or hypersensitive to any of the ingredients;
3. Pneumonia caused by bacteria, mycoplasma, chlamydia, legionella, fungi or other viruses;
4. History of severe chronic respiratory disease and requirement for long-term oxygen therapy
5. Liver disease (such as child Pugh score ≥ grade C, AST more than 5 times of the upper limit of normal
6. Obstructive HABP/VABP induced by lung cancer or other known causes;
7. History of long-term use of immunosuppressive agents;
8. Incapable of understanding study protocol;
9. History of deep venous thrombosis or pulmonary embolism within the last 3 years;
10. Undergoing ECMO or high-frequency oscillatory ventilation support.
11. HIV, hepatitis virus, or syphilis infection;
12. Period of pregnancy or lactation, or planned pregnancy within 6 months;
13. Any condition of unsuitable for the study determined by investigators;
14. Morbid obesity and /or hypertension

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Adverse reaction (AE) and severe AE (SAE) | 28 days
  Safety Assessment
Efficacy Assessment | 28 days
  Time to Clinical Recovery (TTCR)
The Rate of Recovery Without Mechanical Ventilator | 28 days
  Efficacy Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Cetin, Prof, Principal Investigator — TC Erciyes University
Locations (1):
- GENKOK, Kayseri, Melikgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided